CLINICAL TRIAL: NCT00905632
Title: Safety, Antiviral Activity, and Pharmacokinetics of BI 207127 NA Administered in Combination With Peg-IFN and Ribavirin in Chronic HCV-infected Patients for 4 Weeks, a Randomised, Double-blind, Placebo Controlled Study
Brief Title: 4 Week Combination of BI 207127 NA With Peg-IFN and Ribavirin in Chronic HCV Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.7; 2008-008292-34 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — deleobuvir

ARMS (4):
- BI 207127 low dose + SOC (Experimental): BI 207127 low dose tid + SOC
  Interventions: Drug: BI 207127 low dose + SOC
- BI 207127 middle dose +SOC (Experimental): BI 207127 middle dose tid + SOC
  Interventions: Drug: BI 207127 middle dose +SOC
- BI 207127 high dose+SOC (Experimental): BI 207127 high dose tid +SOC
  Interventions: Drug: BI 207127 high dose+SOC
- Placebo + SOC (Placebo Comparator): Placebo tid +SOC
  Interventions: Drug: Placebo + SOC

INTERVENTIONS:
Drug: BI 207127 middle dose +SOC — BI 207127 middle dose tid + SOC
  Arms: BI 207127 middle dose +SOC
Drug: BI 207127 high dose+SOC — BI 207127 high dose tid +SOC
  Arms: BI 207127 high dose+SOC
Drug: Placebo + SOC — Placebo tid +SOC
  Arms: Placebo + SOC
Drug: BI 207127 low dose + SOC — BI 207127 low dose tid + SOC
  Arms: BI 207127 low dose + SOC

SUMMARY:
The main purpose of this clinical trial with BI 207127 is to see the effect of 4 week combination of BI 207127 with Peginterferon alfa (Peg-IFN) and Ribavirin (RBV) on hepatitis C virus (HCV) virus load and how safe BI 207127 is in this combination in HCV infected patients.

ELIGIBILITY:
Inclusion criteria:

1. HCV genotype 1
2. HCV viral load >100,000 IU/mL
3. histology or fibroscan to rule out cirrhosis
4. Absence of retinopathy
5. treatment naive patients and treatment experienced patients
6. Age 18 - 70 years
7. Male OR female with documented hysterectomy OR postmenopausal

Exclusion criteria:

1. Fertile males not willing to use an adequate form of contraception
2. Pretreatment with any HCV-polymerase inhibitor
3. Any concurrent disease if clinically significant based on the investigator's medical assessment
4. Current alcohol or drug abuse, or history of the same
5. Positive test for HIV or HBs
6. History of malignancy
7. Planned or concurrent usage of any other pharmacological therapy including any antiviral therapy or vaccination
8. Usage of any investigational drug within thirty (30) days prior to enrolment or 5 halflives, whichever is longer
9. Any clinically significant laboratory abnormalities based on the investigator's medical assessment at screening
10. Patients treated with any interferon (approved or investigational) or Peg-IFN and/or Ribavirin within 3 months prior to screening
11. Known hypersensitivity to drugs or excipients; Further exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (18):
- France (7):
  - 1241.7.3307A CHU de Grenoble, Grenoble Cédex 9
  - 1241.7.3303A Hôpital Claude Huriez, Lille
  - 1241.7.3302A Hopital de l'Hotel Dieu, Lyon
  - 1241.7.3301A Hôpital Saint Eloi, Montpellier
  - 1241.7.3305A HOP Archet 2, Nice
  - 1241.7.3306A Hôpital Haut-Lévêque, Pessac
  - 1241.7.3304A HOP de Brabois, Vandœuvre-lès-Nancy
- Germany (8):
  - 1241.7.49010 Boehringer Ingelheim Investigational Site, Aachen
  - 1241.7.49012 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.7.49004 Boehringer Ingelheim Investigational Site, Essen
  - 1241.7.49011 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1241.7.49001 Boehringer Ingelheim Investigational Site, Hamburg
  - 1241.7.49013 Boehringer Ingelheim Investigational Site, Mainz
  - 1241.7.49009 Boehringer Ingelheim Investigational Site, Regensburg
  - 1241.7.49002 Boehringer Ingelheim Investigational Site, Ulm
- Switzerland (3):
  - 1241.7.41003 Boehringer Ingelheim Investigational Site, Basel
  - 1241.7.41004 Boehringer Ingelheim Investigational Site, Lugano
  - 1241.7.41001 Boehringer Ingelheim Investigational Site, Sankt Gallen

REFERENCES:
- [Derived] Larrey D, Lohse AW, de Ledinghen V, Trepo C, Gerlach T, Zarski JP, Tran A, Mathurin P, Thimme R, Arasteh K, Trautwein C, Cerny A, Dikopoulos N, Schuchmann M, Heim MH, Gerken G, Stern JO, Wu K, Abdallah N, Girlich B, Scherer J, Berger F, Marquis M, Kukolj G, Bocher W, Steffgen J. Rapid and strong antiviral activity of the non-nucleosidic NS5B polymerase inhibitor BI 207127 in combination with peginterferon alfa 2a and ribavirin. J Hepatol. 2012 Jul;57(1):39-46. doi: 10.1016/j.jhep.2012.02.015. Epub 2012 Mar 10. PMID 22414766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 75 patients were screened, however only 57 patients were randomised.
Groups:
- Treatment Naive (TN): Placebo: Treatment Naive (TN) patients to receive Placebo (given as a tablet, orally three times daily (tid)) + Peg-IFN (Peginterferon alfa (Peg-IFN) injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Naive (TN): BI 207127 400 mg: TN patients to receive 400mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Naive (TN): BI 207127 600 mg: TN patients to receive 600mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Naive (TN): BI 207127 800 mg: TN patients to receive 800mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Experienced (TE): BI 207127 400 mg: Treatment Experienced (TE) patients to receive 400mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Experienced (TE): BI 207127 600 mg: TE patients to receive 600mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
- Treatment Experienced (TE): BI 207127 800 mg: TE patients to receive 800mg BI 207127 NA (given as a tablet, orally three times daily (tid)) + Peg-IFN (injection, sub-cutaneously once a week) + Ribavirin (tablet, orally twice daily (bid)) for 28 days
Period: Overall Study
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Started | 8 | 6 | 7 | 6 | 10 | 9 | 11
Completed | 8 | 6 | 7 | 6 | 10 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who received at least one dose of study medication
Groups:
- Placebo: Patients to receive Placebo + Peg-IFN + Ribavirin tid for 28 days
- Treatment Naive (TN): BI 207127 400 mg: TN patients to receive 400mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Treatment Naive (TN): BI 207127 600 mg: TN patients to receive 600mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Treatment Naive (TN): BI 207127 800 mg: TN patients to receive 800mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Treatment Experienced (TE): BI 207127 400 mg: TE patients to receive 400mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Treatment Experienced (TE): BI 207127 600 mg: TE patients to receive 600mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Treatment Experienced (TE): BI 207127 800 mg: TE patients to receive 800mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg | Total
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.250 (7.573) | 43.833 (15.459) | 42.571 (11.731) | 46.167 (13.963) | 49.200 (5.996) | 50.889 (11.252) | 53.727 (10.287) | 48.930 (10.863)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 0 | 2 | 2 | 10
  Male | 7 | 4 | 5 | 5 | 10 | 7 | 9 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Response Defined as >= 3 Log Drop in Viral Load From Baseline at Day 28 With no Evidence of Virologic Rebound During These 28 Days. Virologic Rebound is Defined as >= 1 Log Increase in Viral Load From Nadir.
Description: The primary efficacy endpoint is the number of participants with virologic response defined as >= 3 log drop in viral load from baseline at day 28 with no evidence of virologic rebound during these 28 days. Virologic rebound is defined as >= 1 log increase in viral load from nadir.
Time Frame: Baseline and 4 weeks
Population: Full Analysis Set (FAS): The subset of patients in the treated set (TS) that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Groups:
- Treatment Naive (TN): Placebo: TN patients to receive Placebo + Peg-IFN + Ribavirin tid for 28 days
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants | 1 | 5 | 7 | 6 | 4 | 5 | 6

2. Secondary Outcome: Viral Load (Log10) at Each Visit up to Day 28, Change From Baseline
Description: Reductions of viral load (Log10) at each visit up to day 28, change from baseline. Change from baseline was calculated as the value at baseline minus the value at each later visit.
  A negative value represents an increase in viral load, a positive value represents a decrease in viral load.
Time Frame: Baseline and days 1, 2, 4, 8, 15, 22 and 28
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy and available viral load data at baseline and day 28.
Measure: Median (Full Range); unit: IU/mL
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 5 | 7 | 6 | 10 | 9 | 11
IU/mL
  Day 1 (02:00 hours) (N=8,5,7,6,10,9,11) | -0.04 [-0.27 to 0.14] | -0.09 [-0.13 to 0.03] | -0.01 [-0.26 to 0.37] | -0.06 [-0.19 to 0.08] | 0.02 [-0.15 to 0.15] | 0.04 [-0.13 to 0.16] | 0.03 [-0.25 to 0.25]
  Day 1 (04:00 hours) (N=8,5,7,6,10,9,11) | -0.05 [-0.28 to 0.04] | -0.27 [-0.36 to -0.11] | -0.28 [-0.54 to 0.07] | -0.29 [-0.56 to 0.10] | -0.10 [-0.37 to 0.08] | -0.09 [-0.36 to 0.21] | -0.01 [-0.81 to 0.31]
  Day 1 (05:55 hours) (N=8,5,7,6,10,9,11) | -0.08 [-0.31 to 0.10] | -0.53 [-0.95 to -0.13] | -0.79 [-1.32 to -0.19] | -1.09 [-1.26 to -0.50] | -0.37 [-0.93 to -0.09] | -0.55 [-0.97 to 0.19] | -0.11 [-1.53 to 0.01]
  Day 1 (08:00 hours) (N=8,5,7,6,10,9,11) | -0.07 [-0.51 to 0.18] | -1.04 [-1.52 to -0.49] | -1.30 [-2.09 to -0.54] | -1.72 [-2.12 to -0.51] | -0.69 [-1.66 to -0.16] | -1.00 [-1.77 to -0.03] | -0.46 [-2.07 to -0.01]
  Day 1 (10:00 hours) (N=8,5,7,6,10,9,11) | -0.06 [-0.34 to 0.15] | -1.15 [-2.13 to -0.53] | -1.70 [-2.53 to -0.77] | -1.99 [-2.75 to -1.41] | -0.80 [-1.80 to -0.44] | -1.18 [-2.44 to -0.22] | -0.79 [-2.45 to -0.20]
  Day 1 (11:55 hours) (N=8,5,7,6,10,9,11) | -0.10 [-0.50 to 0.20] | -1.50 [-2.51 to -0.54] | -2.38 [-2.89 to -1.02] | -2.40 [-3.22 to -1.55] | -1.11 [-2.53 to -0.61] | -1.66 [-2.72 to -0.42] | -1.01 [-2.53 to -0.20]
  Day 1 (15:00 hours) (N=8,5,7,6,8,9,10) | -0.20 [-0.49 to 0.05] | -2.13 [-3.05 to -0.71] | -2.49 [-3.36 to -1.30] | -2.86 [-3.52 to -2.48] | -1.45 [-3.02 to -0.92] | -2.48 [-3.05 to -0.66] | -1.66 [-2.79 to -0.78]
  Day 2 (N=8,5,7,6,10,8,11) | -0.39 [-1.02 to 0.24] | -1.78 [-3.86 to -0.60] | -2.73 [-4.07 to -2.18] | -3.32 [-3.90 to -3.17] | -1.57 [-3.54 to -0.46] | -2.46 [-3.55 to -0.87] | -1.93 [-2.98 to -0.62]
  Day 4 (N=8,5,7,6,10,9,11) | -0.61 [-0.93 to 0.04] | -2.43 [-4.33 to -1.43] | -3.07 [-5.25 to -2.95] | -3.80 [-4.11 to -3.52] | -1.51 [-4.15 to -0.54] | -2.76 [-3.92 to -0.92] | -2.53 [-3.54 to -1.19]
  Day 8 (N=8,5,7,6,10,9,9) | -0.32 [-1.43 to 0.26] | -3.19 [-5.28 to -1.83] | -4.13 [-6.36 to -3.28] | -4.31 [-4.95 to -3.77] | -1.58 [-4.86 to -0.36] | -3.04 [-4.51 to -0.88] | -2.68 [-4.08 to -1.90]
  Day 15 (N=7,5,7,6,10,8,8) | -0.42 [-1.50 to -0.11] | -3.89 [-5.74 to -2.96] | -5.27 [-6.36 to -3.86] | -4.86 [-5.20 to -4.45] | -2.09 [-4.96 to -0.70] | -4.00 [-5.60 to -1.37] | -3.26 [-4.68 to -2.11]
  Day 22 (N=8,5,7,6,10,8 ,8) | -1.06 [-2.78 to -0.45] | -4.53 [-5.74 to -3.77] | -5.55 [-6.36 to -4.62] | -5.27 [-5.90 to -4.46] | -2.63 [-4.96 to -1.42] | -3.83 [-5.71 to -1.65] | -4.13 [-4.98 to -2.40]
  Day 28 (N=7,5,6,6,10,8,7) | -1.41 [-3.75 to -0.73] | -5.08 [-5.74 to -4.32] | -5.61 [-6.22 to -4.84] | -5.44 [-5.90 to -4.93] | -2.86 [-4.96 to -1.32] | -4.20 [-6.14 to -1.20] | -4.48 [-5.41 to -2.99]

3. Secondary Outcome: Viral Load at Each Visit up to Day 28
Description: Viral load (VL) (original values) at each visit up to day 28.
Time Frame: Baseline and days 8, 15, 22 and 28
Population: Pharmacodynamic (PD) set which included patients in the treated set but excluded VL values after recorded treatment stop time and values after subjects took wrong or additional doses of treatment. Also one patient was excluded from all descriptive PD summaries due to a protocol violation and another excluded as they did not have a predose VL value.
Measure: Median (Full Range); unit: IU/mL
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
IU/mL
  Baseline (N=8,4,7,6,9,9,11) | 3540000 [925000 to 10900000] | 3260000 [572000 to 4910000] | 8480000 [629000 to 20600000] | 3440000 [763000 to 19000000] | 3620000 [1330000 to 17400000] | 3560000 [684000 to 12300000] | 3340000 [665000 to 45300000]
  Day 8 (N=8,3,6,6,9,9,9) | 1520000 [34500 to 19700000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | 320 [42.0 to 3200] | 234 [28.0 to 913] | 47800 [30 to 2300000] | 4120 [161 to 89400] | 8460 [108 to 566000]
  Day 15 (N=7,2,3,4,8,8,7) | 618000 [92800 to 6470000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | 107 [28.0 to 188] | 18100 [367 to 626000] | 690 [31 to 153000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data.
  Day 22 (N=8,1,2,2,8,5,6) | 249000 [1550 to 3870000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | 29600 [554 to 70400] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data.
  Day 28 (N=7,1,2,0,7,5,4) | 168000 [133 to 1620000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No patients with available data at this timepoint. | 43100 [685 to 373000] | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data. | NA [NA to NA] — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 of subjects had detectable data.

4. Secondary Outcome: Number of Participants With Virologic Response at Day 28
Description: Number of participants with virologic response at day 28, defined as achieving viral load below the limit of quantification (BLQ), <10 IU/mL, at day 28
Time Frame: day 28
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants | 0 | 4 | 6 | 6 | 1 | 3 | 2

5. Secondary Outcome: Number of Participants With Rapid Virological Response
Description: Number of participants with rapid virological response - defined as serum Hepatitis C virus (HCV) RNA level below the limit of detection (BLD) of the Roche COBAS Taqman HCV/High Pure System (HPS) for extraction assay (10 IU/mL) on Day 28.
Time Frame: 4 weeks
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants | 0 | 3 | 4 | 3 | 0 | 2 | 2

6. Secondary Outcome: Number of Participants With Early Virological Response
Description: Number of participants with early virological response (EVR) defined as at least 2log10 reduction in HCV Ribonucleic acid (RNA) from baseline at Week 12. Number of responders* - Response = At least a 2 log10 reduction in viral load from baseline at Week 12 (Day 84)
Time Frame: Baseline and week 12
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants
  Number of responders | 7 | 5 | 7 | 6 | 6 | 6 | 4
  Number of failures | 1 | 1 | 0 | 0 | 4 | 3 | 7

7. Secondary Outcome: Number of Participants With End of Treatment Response
Description: Number of participants with end of treatment response (ETR) - defined as serum HCV RNA level below the limit of detection (BLD) of the Roche COBAS Taqman HCV/HPS assay (10 IU/mL) at end of treatment (including 5-day washout). Number of responders* - Response = Viral load below the limit of detection at end of all treatment.
Time Frame: Week 12
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants
  Number of responders | 4 | 3 | 6 | 6 | 4 | 3 | 1
  Number of failures | 4 | 3 | 1 | 0 | 6 | 6 | 10

8. Secondary Outcome: Number of Participants With Sustained Virological Response
Description: Number of participants with sustained virological response. Sustained virological response was defined as serum HCV RNA below the limit of detection (<10 IU/mL) at least 85 days after stopping standard care (SOC).
Time Frame: Until end of treatment, up to 570 days
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: Participants
Arm/Group | Treatment Naive (TN): Placebo | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 8 | 6 | 7 | 6 | 10 | 9 | 11
Participants
  Number of responders | 2 | 2 | 5 | 6 | 0 | 0 | 0
  Number of failures | 6 | 4 | 2 | 0 | 10 | 9 | 11

9. Secondary Outcome: Plasma Concentration Time Profiles of BI 207127
Description: Plasma concentration time profiles of BI 207127
Time Frame: 0.5 hours (h), 3h, 8h, 15h, 23.917h, 503.917h, 649h, 652h, 656h and 672h after drug administration
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy. One patient in the TE: BI 207127 400 mg group was excluded from the analysis due to a protocol violation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 9 | 11
ng/mL
  BI 207127 0.5 hours (N=4,6,6,-,8,-) | 111 (344) | 103 (534) | 230 (391) | NA (NA) — Some patients had data below the limit of quantification which is not analysable and per internal rules, descriptive statistics are not calculated unless data from at least 2/3rds of all subjects were available. | 422 (265) | NA (NA) — Some patients had data below the limit of quantification which is not analysable and per internal rules, descriptive statistics are not calculated unless data from at least 2/3rds of all subjects were available.
  BI 207127 3 hours (N=6,7,6,9,9,10) | 2040 (32.4) | 2610 (76.0) | 5730 (52.4) | 3070 (64.3) | 4650 (90.4) | 4460 (59.8)
  BI 207127 8 hours (N=6,7,6,9,9,11) | 2590 (29.0) | 4610 (124) | 12600 (65.3) | 4320 (81.1) | 6070 (67.3) | 7140 (73.1)
  BI 207127 15 hours (N=6,7,6,8,9,10) | 3550 (55.3) | 6530 (55.9) | 13500 (62.8) | 4860 (115) | 7270 (93.4) | 13300 (67.2)
  BI 207127 23.917 hours (N=6,7,6,9,8,11) | 595 (72.0) | 1610 (138) | 4780 (76.4) | 1170 (201) | 3450 (173) | 9350 (71.0)
  BI 207127 503.917 hours (N=6,7,5,9,8,8) | 336 (101) | 1250 (302) | 1730 (146) | 330 (104) | 709 (167) | 4460 (249)
  BI 207127 649 hours (N=6,7,6,9,8,7) | 1210 (91.4) | 2490 (176) | 2340 (197) | 1050 (100) | 1710 (153) | 3050 (182)
  BI 207127 652 hours (N=6,7,6,9,8,7) | 2520 (86.3) | 5100 (100) | 11300 (68.6) | 2650 (66.3) | 5340 (60.0) | 9070 (106)
  BI 207127 656 hours (N=5,7,6,8,8,6) | 905 (113) | 1940 (121) | 2820 (145) | 635 (82.7) | 1380 (97.5) | 3820 (122)
  BI 207127 672 hours (N=5,7,6,-,8,6) | 57.7 (137) | 80.4 (306) | 101 (175) | NA (NA) — Some patients had data below the limit of quantification which is not analysable and per internal rules, descriptive statistics are not calculated unless data from at least 2/3rds of all subjects were available. | 62.4 (105) | 163 (236)

10. Secondary Outcome: Plasma Concentration Time Profiles of CD 6168
Description: Plasma concentration time profiles of CD 6168
Time Frame: 0.5 hours (h), 3h, 8h, 15h, 23.917h, 503.917h, 649h, 652h, 656h and 672h after drug administration
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 9 | 11
ng/mL
  CD 6168 0.5 hours (N=-,-,-,-,-,-) | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification. | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification. | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification. | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification. | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification. | NA (NA) — No descriptive statistics calculated as all participants results were below the limit of quantification.
  CD 6168 3 hours (N=6,7,6,9,8,11) | 124 (152) | 155 (68.1) | 397 (47.6) | 142 (63.4) | 247 (58.1) | 183 (144)
  CD 6168 8 hours (N=6,7,6,9,9,11) | 337 (61.6) | 636 (97.3) | 1220 (39.0) | 307 (79.1) | 545 (64.1) | 622 (54.8)
  CD 6168 15 hours (N=6,7,5,8,9,10) | 690 (57.8) | 1320 (55.2) | 2210 (47.0) | 570 (122) | 973 (64.6) | 1330 (61.9)
  CD 6168 23.917 hours (N=6,7,6,9,8,11) | 201 (71.7) | 617 (136) | 1530 (57.3) | 276 (186) | 827 (143) | 1920 (55.2)
  CD 6168 503.917 hours (N=6,7,5,9,8,8) | 193 (89.4) | 712 (308) | 1310 (218) | 150 (164) | 385 (123) | 2730 (285)
  CD 6168 649 hours (N=6,7,6,9,8,7) | 394 (89.4) | 1230 (193) | 1160 (234) | 196 (169) | 473 (132) | 1470 (249)
  CD 6168 652 hours (N=6,7,6,9,8,7) | 699 (53.9) | 1940 (144) | 3360 (105) | 556 (104) | 1160 (71.8) | 2570 (207)
  CD 6168 656 hours (N=5,7,6,8,8,6) | 418 (81.4) | 1200 (153) | 1660 (194) | 243 (135) | 566 (106) | 1770 (178)
  CD 6168 672 hours (N=4,7,5,-,6,6) | 61.7 (58.8) | 84.8 (490) | 135 (337) | NA (NA) — Some patients had data below the limit of quantification which is not analysable and per internal rules, descriptive statistics are not calculated unless data from at least 2/3rds of all subjects were available. | 50.8 (90.8) | 123 (297)

11. Secondary Outcome: Cmax of BI 207127 and CD 6168 in Plasma After First Dose and After Last Dose (Steady State)
Description: Maximum measured concentration of the analyte in plasma (Cmax) after first dose on day 1 (Cmax) and after last dose (steady state) on day 28 (Cmax,ss) of BI 207127 and CD 6168
Time Frame: 5 min before drug admin and 30min, 1 hour (h), 2h, 3h, 4h, 5h 55min, 8h, 10h, 11h 55min and 15h after drug administration on day 1: 5 min before drug admin and 30min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 48h after admin on day 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 9 | 11
ng/mL
  Cmax BI207127 in plasma (N=6,7,6,9,9,11) | 2420 (29.1) | 3490 (61.7) | 7440 (81.8) | 3590 (64.1) | 5910 (54.3) | 7640 (52.5)
  Cmax CD 6168 in plasma (N=6,7,6,9,8,11) | 261 (56.2) | 412 (64.5) | 891 (51.0) | 232 (69.4) | 426 (75.5) | 556 (75.7)
  Cmax,ss BI207127 in plasma (N=6,7,6,9,9,7) | 3260 (70.1) | 6020 (91.5) | 12200 (73.0) | 3460 (55.2) | 5750 (67.2) | 10800 (66.0)
  Cmax,ss CD 6168 in plasma (N=6,7,6,9,8,7) | 861 (36.0) | 2090 (135) | 3450 (107) | 584 (105) | 1170 (74.0) | 2990 (122)

12. Secondary Outcome: Tmax of BI 207127 and CD 6168 in Plasma After First Dose and After Last Dose (Steady State)
Description: tmax [h] Time from (last) dosing to the maximum measured concentration of the analyte in plasma after first dose on day 1 and after last dose on day 28 (steady state).
Time Frame: as for outcome 11
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 9 | 11
hour
  tmax BI 207127 (N=6,7,6,9,9,11) | 2.96 (27.8) | 3.87 (24.4) | 3.91 (24.9) | 3.11 (29.1) | 3.19 (31.7) | 4.10 (83.1)
  tmax CD 6168 (N=6,7,6,9,9,11) | 4.79 (27.9) | 4.80 (28.2) | 5.56 (16.3) | 4.82 (26.1) | 5.69 (13.4) | 5.37 (23.0)
  tmax,ss BI 207127 (N=6,7,6,9,8,7) | 2.57 (108) | 3.56 (41.0) | 3.32 (16.5) | 2.77 (27.4) | 3.26 (24.5) | 3.91 (23.3)
  tmax,ss CD 6168(N=6,7,6,9,8,7) | 3.24 (68.0) | 4.34 (32.0) | 3.91 (24.0) | 3.85 (27.5) | 3.63 (24.6) | 3.49 (62.1)

13. Secondary Outcome: AUC0-6 of BI 207127 and CD 6168 in Plasma After First Dose and After Last Dose (Steady State)
Description: Area under the concentration-time curve of the analyte in plasma (AUC) after first dose on day 1 (AUC0-6) and after last dose on day 28 (AUC0-6,ss) of BI 207127 and CD 6168
Time Frame: 30min, 1 hour (h), 2h, 3h, 4h and 5h 55min after drug administration on day 1: 30min, 1h, 2h, 3h, 4h and 6h after admin on day 28
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 5 | 5 | 5 | 9 | 9 | 7
ng*h/mL
  AUC0-6 BI 207127 (N=5,5,5,9,9,7) | 8840 (35.0) | 13500 (61.5) | 23700 (62.6) | 13000 (64.8) | 21900 (70.3) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.
  AUC0-6 CD 6168 (N=-,-,-,-,-,-) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.
  AUC0-6,ss BI 207127 (N=6,7,7,8,8,7) | 11300 (83.7) | 24000 (112) | 42500 (88.1) | 12400 (56.1) | 21400 (73.7) | 36600 (107)
  AUC0-6,ss CD 6168 (N=6,7,7,9,8,7) | 3180 (48.7) | 9610 (162) | 14000 (138) | 2380 (115) | 4920 (90.2) | 12500 (191)

14. Secondary Outcome: Cpre Pharmacokinetic Parameter of BI 207127 and CD 6168
Description: Cpre,N [ng/mL] - Predose concentration of the analyte in plasma immediately before administration of the Nth dose after N-1 doses were administered for BI 207127 and CD 6168. Descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. All values for Cpre,1 were not available, therefore no results are presented below.
Time Frame: 5 minutes before drug administration on days 1, 2, 4, 8, 15, 22 and 27
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 9 | 11
ng/mL
  BI 207127 Cpre,1 (N=-,-,-,-,-,-) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.
  BI 207127 Cpre,2 (N=6,7,6,9,8,11) | 595 (72.0) | 1610 (138) | 4780 (76.4) | 1170 (201) | 3450 (173) | 9350 (71.0)
  BI 207127 Cpre,4 (N=5,6,6,9,9,10) | 659 (48.4) | 1530 (267) | 6200 (160) | 816 (197) | 2780 (201) | 9830 (170)
  BI 207127 Cpre,8 (N=6,6,5,9,9,9) | 414 (117) | 607 (131) | 1770 (310) | 635 (217) | 783 (186) | 4160 (176)
  BI 207127 Cpre,15 (N=6,7,6,9,8,8) | 399 (135) | 1170 (188) | 1560 (139) | 358 (97.8) | 944 (163) | 3530 (349)
  BI 207127 Cpre,22 (N=6,7,6,9,8,8) | 336 (101) | 1250 (302) | 1340 (165) | 330 (104) | 709 (167) | 4460 (249)
  BI 207127 Cpre,27 (N=-,5,-,6,-,-) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | 4270 (56.9) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | 1280 (80.8) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.
  CD 6168 Cpre,1 (N=-,-,-,-,-,-) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.
  CD 6168 Cpre,2 (N=6,7,6,9,8,11) | 201 (71.7) | 617 (136) | 1530 (57.3) | 276 (186) | 827 (143) | 1920 (55.2)
  CD 6168 Cpre,4 (N=5,6,6,9,9,10) | 236 (56.2) | 564 (276) | 2510 (146) | 250 (257) | 994 (192) | 3000 (235)
  CD 6168 Cpre,8 (N=6,6,5,9,9,9) | 194 (111) | 368 (138) | 1140 (177) | 253 (353) | 350 (221) | 2340 (183)
  CD 6168 Cpre,15 (N=6,7,6,9,8,8) | 239 (175) | 723 (265) | 1000 (149) | 169 (172) | 428 (135) | 2020 (519)
  CD 6168 Cpre,22 (N=6,7,6,9,8,8) | 193 (89.4) | 712 (308) | 1010 (226) | 150 (164) | 385 (123) | 2730 (285)
  CD 6168 Cpre,27 (N=-,5,-,6,-,-) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | 1730 (74.5) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | 427 (147) | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available. | NA (NA) — No descriptive statistics calculated. Per internal rules descriptive statistics were calculated only if at least 2/3 plasma concentrations were available.

15. Secondary Outcome: C6,ss Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State After the Last Dose
Description: C6,ss Pharmacokinetic parameters of BI 207127 and CD 6168 at steady state after the last dose. C6,ss is the concentration 6 hours after dosing at steady-state (reported as 654 h).
Time Frame: 654 hours after drug administration on day 28
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy and available endpoint data at day 28. One patient in the TE: BI 207127 400 mg group was excluded from the analysis due to a protocol violation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 8 | 7
ng/mL
  BI 207127 654 hours | 1520 (103) | 4030 (107) | 5820 (94.4) | 1380 (71.4) | 2810 (85.7) | 5910 (114)
  CD 6168 654 hours | 556 (63.7) | 1810 (148) | 2580 (136) | 424 (122) | 893 (89.7) | 2200 (133)

16. Secondary Outcome: AUC0-infinity,ss Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State After the Last Dose
Description: Area under the concentration time curve of the analyte in plasma over the time interval of 0 to infinity at steady state (AUC0-infinity,ss): Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State (SS) After the Last Dose
Time Frame: 5 min before drug admin and 30min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 48h after admin on day 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 8 | 8 | 6
ng*h/mL
  AUC0 to infinity,SS of BI207127 | 20500 (88.4) | 38600 (131) | 62300 (99.2) | 16900 (63.0) | 31500 (79.2) | 71300 (116)
  AUC0 to infinity,SS of CD 6168 | 7170 (70.9) | 19600 (201) | 26800 (171) | 4290 (129) | 9190 (97.9) | 29000 (196)

17. Secondary Outcome: λz Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State After the Last Dose
Description: Terminal rate constant in plasma (λz): Pharmacokinetic parameters of BI 207127 and CD 6168 at steady state after the last dose
Time Frame: 5 min before drug admin and 30min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 48h after admin on day 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 8 | 8 | 6
1/h
  λz,ss of BI 207127 | 0.162 (17.6) | 0.182 (27.8) | 0.170 (32.6) | 0.226 (20.8) | 0.163 (30.9) | 0.174 (28.2)
  λz,ss of CD 6168 | 0.157 (36.4) | 0.163 (20.3) | 0.166 (43.3) | 0.185 (21.4) | 0.192 (24.3) | 0.129 (56.0)

18. Secondary Outcome: t1/2,ss and MRTpo,ss Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State After the Last Dose
Description: Terminal half-life of the analyte in plasma at steady state (t1/2,ss) and mean residence time of the analyte in the body at steady state after oral administration (MRTpo,ss): Pharmacokinetic parameters of BI 207127 and CD 6168 at steady state after the last dose
Time Frame: 5 min before drug admin and 30min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 48h after admin on day 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 5 | 7 | 6 | 8 | 8 | 6
hour
  t1/2,ss of BI 207127 | 4.28 (17.6) | 3.81 (27.8) | 4.09 (32.6) | 3.06 (20.8) | 4.26 (30.9) | 3.99 (28.2)
  MRTpo,ss of BI 207127 | 6.44 (28.3) | 6.40 (17.7) | 5.83 (14.5) | 5.32 (16.8) | 5.82 (12.9) | 7.03 (23.8)
  t1/2,ss of CD 6168 | 4.42 (36.4) | 4.25 (20.3) | 4.18 (43.3) | 3.75 (21.4) | 3.61 (24.3) | 5.36 (56.0)
  MRTpo,ss of CD 6168 | 8.98 (26.0) | 8.61 (24.7) | 8.07 (22.5) | 7.51 (14.2) | 7.75 (16.4) | 9.38 (30.8)

19. Secondary Outcome: RA,Cmax Pharmacokinetic Parameters of BI 207127 and CD 6168 at Steady State After the Last Dose
Description: Accumulation ratio of maximum measured concentration of the analyte in plasma (RA,Cmax): Pharmacokinetic parameters of BI 207127 and CD 6168 at steady state after the last dose. Ratio was calculated as Cmax,ss divided by Cmax.
Time Frame: 5 min before drug admin and 30min, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h and 48h after admin on day 28
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Treatment Naive (TN): BI 207127 400 mg | Treatment Naive (TN): BI 207127 600 mg | Treatment Naive (TN): BI 207127 800 mg | Treatment Experienced (TE): BI 207127 400 mg | Treatment Experienced (TE): BI 207127 600 mg | Treatment Experienced (TE): BI 207127 800 mg
Number analyzed (Participants) | 6 | 7 | 6 | 9 | 8 | 7
ratio
  RA,Cmax of BI 207127 | 1.35 (74.1) | 1.72 (95.2) | 1.64 (84.4) | 0.965 (37.5) | 1.02 (40.0) | 1.44 (56.2)
  RA,Cmax of CD 6168 | 3.30 (66.5) | 5.07 (127) | 3.87 (120) | 2.52 (84.8) | 2.77 (55.9) | 6.08 (146)

20. Secondary Outcome: Number of Participants With Clinical Relevant Abnormalities for Vital Signs, Body Temperature, Physical Examination, Blood Chemistry, Haematology, Coagulation, Urinalysis and ECG
Description: Number of participants with clinically relevant abnormalities for vital signs, blood chemistry, body temperature, physical examination, haematology, coagulation, urinalysis and electrocardiography (ECG). New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: From the start of the study to Day 30 (2 days after last dose)
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: participants
Groups:
- BI 207127 400 mg: Patients to receive 400mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- BI 207127 600 mg: Patients to receive 600mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
- BI 207127 800 mg: Patients to receive 800mg BI 207127 NA tablet + Peg-IFN + Ribavirin tid for 28 days
Arm/Group | Placebo | BI 207127 400 mg | BI 207127 600 mg | BI 207127 800 mg
Number analyzed (Participants) | 8 | 16 | 16 | 17
participants
  Weight decreased | 0 | 0 | 1 | 3
  Alanine aminotransferase increased | 0 | 1 | 2 | 1

21. Secondary Outcome: Number of Participants With Discontinuations Due to AEs
Description: Number of participants with adverse events (AEs) leading to discontinuation of trial drug
Time Frame: 4 weeks
Population: Full Analysis Set (FAS): The subset of patients in the TS that had at least one measurement of efficacy.
Measure: Number; unit: participants
Arm/Group | Placebo | BI 207127 400 mg | BI 207127 600 mg | BI 207127 800 mg
Number analyzed (Participants) | 8 | 16 | 16 | 17
participants | 0 | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: From drug administration until 2 days after the end of treatment, up to 570 days
Arm/Group | Placebo | BI 207127 400 mg | BI 207127 600 mg | BI 207127 800 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 2/16 | 0/16 | 1/17
Other Adverse Events (participants affected / at risk) | 7/8 | 16/16 | 16/16 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | BI 207127 400 mg (N=16) | BI 207127 600 mg (N=16) | BI 207127 800 mg (N=17)
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | BI 207127 400 mg (N=16) | BI 207127 600 mg (N=16) | BI 207127 800 mg (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 10 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 4 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 4 | 6 | 9
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 8
Asthenia (General disorders) | 1 | 7 | 5 | 4
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 3 | 0
Fatigue (General disorders) | 2 | 2 | 5 | 5
Feeling cold (General disorders) | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 8 | 2 | 4
Injection site erythema (General disorders) | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 1 | 0 | 0 | 1
Irritability (General disorders) | 2 | 4 | 1 | 2
Malaise (General disorders) | 0 | 1 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 1
General physical condition normal (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4 | 9
Hyperphagia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Growing pains (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 6 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 4
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 2
Formication (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 6 | 7 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 4
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 6 | 5
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2 | 0 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Breast discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BIs intellectual property rights.